CLINICAL TRIAL: NCT00118300
Title: Phase I Study of Capecitabine (Xeloda) and Radiation Therapy in Patients With Locally Advanced Cervical and Pelvic Malignancies
Brief Title: Capecitabine and Radiation Therapy in Treating Patients With Locally Advanced Cervical Cancer or Other Pelvic Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Competing studies
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Charles Kunos, MD, PhD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE9804; P30CA043703 (NIH); CASE-9804 (Other: Case Comphrensive Cancer Center); CWRU-010514
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-07

CONDITIONS: Cervical Cancer; Endometrial Cancer; Ovarian Cancer; Vaginal Cancer
Keywords: stage III cervical cancer; stage IVA cervical cancer; recurrent cervical cancer; stage III endometrial carcinoma; recurrent endometrial carcinoma; stage III ovarian epithelial cancer; recurrent ovarian epithelial cancer; stage III ovarian germ cell tumor; recurrent ovarian germ cell tumor; stage III vaginal cancer; stage IVA vaginal cancer; recurrent vaginal cancer; ovarian sarcoma; ovarian stromal cancer; stage IV endometrial carcinoma; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage II vaginal cancer; stage I vaginal cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Vaginal Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Capecitabine; Brachytherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine — Patients also receive oral capecitabine twice daily 7 days a week in weeks 1-5 and 7-8. Courses repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.
Radiation: brachytherapy — 1 or 2 applications of low-dose rate intracavitary brachytherapy in weeks 7-8 OR 5 applications of high-dose rate (HDR)* intracavitary brachytherapy once weekly in weeks 4-8.
Radiation: radiation therapy — Patients undergo external beam radiotherapy to the whole pelvis once daily 5 days a week in weeks 1-5.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. Giving chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of capecitabine when given together with radiation therapy in treating patients with locally advanced cervical cancer or other pelvic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and dose-limiting toxicity of capecitabine when given in combination with pelvic external beam radiotherapy and intracavitary brachytherapy in patients with primary or recurrent locally advanced cervical cancer or other pelvic malignancy.

Secondary

* Determine the clinical anti-tumor response in patients treated with this regimen.
* Determine adverse clinical sequelae in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of capecitabine.

Patients undergo external beam radiotherapy to the whole pelvis once daily 5 days a week in weeks 1-5 and receive 1 or 2 applications of low-dose rate intracavitary brachytherapy in weeks 7-8 OR 5 applications of high-dose rate (HDR)* intracavitary brachytherapy once weekly in weeks 4-8. Patients also receive oral capecitabine twice daily 7 days a week in weeks 1-5 and 7-8. Courses repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.

NOTE: *No external beam radiotherapy is administered on the day of HDR brachytherapy. If the majority of external beam radiotherapy has been administered, HDR brachytherapy may be administered in 2 applications per week (separated by at least 72 hours) in order to complete all treatment by week 8.

Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A minimum of 6 patients are treated at the MTD.

After completion of study treatment, patients are followed at 1 month, every 3 months for 1 year, every 6 months for 2 years, and then annually for 2 years.

PROJECTED ACCRUAL: Approximately 4-24 patients will be accrued for this study within 2-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cervical cancer or other pelvic malignancy, including vaginal, endometrial, or ovarian cancer

  * Primary or recurrent disease
  * Locally advanced disease, defined as the following:

    * Stage IB2-IVA (for cervical or vaginal cancer)
    * Any non-extra pelvic metastatic stage (for endometrial or ovarian cancer)
* Not amenable to curative surgical resection alone
* Bidimensionally measurable or clinically evaluable disease
* Refused or ineligible for weekly IV cisplatin chemotherapy due to renal insufficiency, prior platinum adverse sensitivity, pre-existing neuropathy, or concurrent co-morbid illness
* No histologically confirmed or clinically suspicious (≥ 1 cm) para-aortic lymphadenopathy
* No brain metastases or primary brain tumors

PATIENT CHARACTERISTICS:

Age

* 18 and over (80 and under for second and third dose-escalation levels)

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* AST and ALT < 2 times upper limit of normal

Renal

* See Disease Characteristics
* Creatinine normal OR
* Creatinine clearance ≥ 30 mL/min*
* No proteinuria or clinically significant impaired renal function NOTE: *Creatine clearance testing required in patients > 60 years of age

Cardiovascular

* No symptomatic New York Heart Association class III or IV congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No uncontrolled hypertension

Gastrointestinal

* Able to swallow oral medication
* No bowel obstruction
* No malabsorption illness

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known hypersensitivity to capecitabine or fluorouracil
* No ongoing or active infection
* No other uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No other active invasive malignancy

  * Prior malignancy in remission for ≥ 6 months that is not currently being treated allowed

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Recovered from prior chemotherapy
* At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas)
* Prior chemotherapy for a non-gynecologic malignancy or in the adjuvant setting allowed
* No prior capecitabine

Endocrine therapy

* Prior adjuvant hormonal therapy allowed

Radiotherapy

* Recovered from prior radiotherapy
* At least 4 weeks since prior radiotherapy
* Prior radiotherapy for a non-gynecologic malignancy allowed
* No prior low abdominal or pelvic radiotherapy

Surgery

* Not specified

Other

* At least 3 weeks since prior investigational anticancer agents and recovered
* No prior anticancer treatment that contraindicates study therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-04

PRIMARY OUTCOMES:
Maximum tolerated dose | weekly
Disease response measured prior to brachytherapy and at 1 month after completion of study treatment | 1 month after completion of study treatment
Toxicity as measured by CTC v 3.0 weekly | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kunos, MD, PhD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/results?term=case9804